CLINICAL TRIAL: NCT05157178
Title: Immunogenicity Study of the Covid-19 (Recombinante) Vaccine - Fiocruz/AstraZeneca When Administered With a 4 or 8 Weeks Interval Between the First Two Doses.
Brief Title: Immunogenicity Study of the Covid-19 (Recombinante) Vaccine With a 4 or 8 Week Interval Between the First Doses.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ASCLIN 004/2021
Record Dates: First submitted 2021-12-10; First posted 2021-12-14 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Vaccines

STUDY DESIGN:
Masking Description: Only the laboratory technician is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 4 week interval (Experimental): Administration of two doses of the Covid-19 (recombinante) vaccine, with a 4 week interval between the two doses.
  Interventions: Biological: Covid-19 (recombinante) vaccine
- 8 week interval (Experimental): Administration of two doses of the Covid-19 (recombinante) vaccine, with a 8 week interval between the two doses.
  Interventions: Biological: Covid-19 (recombinante) vaccine
- 12 week interval (Active Comparator): Administration of two doses of the Covid-19 (recombinante) vaccine, with a 12 week interval between the two doses.
  Interventions: Biological: Covid-19 (recombinante) vaccine

INTERVENTIONS:
Biological: Covid-19 (recombinante) vaccine — Administration of the Covid-19 (recombinante) vaccine

SUMMARY:
The purpose of this clinical trial is to compare antibody response and safety of the Covid-19 (recombinante) vaccine according to different time intervals between the first two doses (4, 8 and 12 weeks) and serologic status immediately before the vaccine.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants giving written informed consent will be evaluated for eligibility criteria. At day 0, participants who meet the eligibility requirements will undergo a thorough medical evaluation and a urine pregnancy test (if applicable). Eligible participants will be placed in one of three vaccination interval groups (4, 8 or 12 weeks between the first two Covid -19 (recombinante) vaccine doses) in a randomized manner, via a computer program created by the statistical annalist. Both participant and research team will know the allocated group.

Eligible and consenting participants will have a blood sample collected (IgG Anti-S antibodies) and immediately after be administered a third dose of the Covid-19 (recombinante) vaccine. Participants will be instructed to fill out an adverse events journal for solicited adverse events for 7 days and non-solicited adverse events for 28 days after each dose. The research team will contact the participant remotely at least twice during the first two weeks.

The participant will return for a follow-up visit to the research center 28 days after each dose, to evaluate adverse events, collect blood samples (IgG Anti-S antibodies) and undergo a thorough medical evaluation.

The participant will also return to the research center to collect blood samples (IgG Anti-S antibodies) in two more follow-up visits: 6 and 12 months after vaccination with Covid-19 (recombinante).

ELIGIBILITY:
Inclusion Criteria:

* Availability to participate during the entire study, and ability to follow study protocol strictly.
* Consent to supply personal contact information, such as telephone numbers, address and other information so the research team may contact the participant (For example, in case the participant fails to attend a scheduled visit without previous notice)
* Ability to understand and sign the volunteered and informed consent form, and ability to fill in the adverse events journal at home, according to the evaluation of the principal investigator ou delegated research team members.
* Understanding the impossibility of participating in another clinical trial while participating in this clinical trial.
* Ability to fill out the adverse events journal at home

Exclusion Criteria:

* Pregnancy or puerperium
* Having received any other Covid-19 vaccine any time before inclusion in the study
* Having received any other vaccine 30 days before inclusion in the study
* Covid-19 disease confirmed by RT-PCR (Real time polymerase chain reaction) up to 28 days before inclusion in the study.
* Covid-19 symptoms during evaluation of inclusion in the study (Day 0).
* Fever (Axillary temperature above 37,8 º C / 100,04 °F) 72 hours before vaccination in the study.
* Contraindications to the Covid-19 (recombinante) vaccine - Fiocruz/AstraZeneca
* Use of immunosuppressive medication, such as systemic corticosteroids or chemotherapy, or immunosuppressive diseases. We will consider as immunosuppressive doses of systemic corticosteroids daily doses of prednisone of 10mg or more, for more than 14 days.
* Any discoveries made by the principal investigator that would enhance the risk of an adverse result following the participation in the study, or that in some other way justifies exclusion from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1264 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titers of IgG Anti-S antibody after two doses of Covid-19 (recombinante) | 6 months
  Geometric mean titers of IgG Anti-S antibodies, obtained immediately before the first dose and 28 days after the second dose of the Covid-19 (recombinante) vaccine, comparing 4 and 8 week intervals to 12 weeks interval between the first two to doses

SECONDARY OUTCOMES:
Seroconversion of IgG Anti-S antibodies after two doses of Covid-19 (recombinante) vaccination | 6 months
  Seroconversion proportion, defined by an elevation of Anti-S antibody titers four times after two doses of Covid-19 (recombinante), in comparison to baseline (immediately before the first dose), comparing 4 and 8 week intervals to 12 weeks interval between the first two to doses
Seroconversion of IgG Anti-S antibodies after two doses of Covid-19 (recombinante) by serologic status before vaccination | 6 months
  Seroconversion proportion, defined by an elevation of Anti-S antibody titers four times after two doses of Covid-19 (recombinante), in comparison to baseline (immediately before the first dose), comparing 4 and 8 week intervals to 12 weeks interval between the first two to doses and serologic status before vaccination
Geometric mean titer of Anti-S IgG antibodies 6 and 12 months after Covid-19 (recombinante) vaccination | 15 months
  Geometric mean titer of Anti-S IgG antibodies 6 and 12 months after the vaccination, according to vaccination interval group (4, 8 ans 12 weeks) and serologic status before vaccination.
Reactogenicity and Safety of Covid-19 (recombinante) vaccine | 15 months
  Frequency, intensity and causality of solicited and non solicited adverse events up to 28 days after vaccination with Covid-19 (recombinante) vaccine. Frequency and causality of severe adverse events throughout participation in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Clarice Monteiro Vianna, Principal Investigator — Bio-Manguinhos/Fiocruz
Locations (4):
- Brazil (4):
  - Instituto de Tecnologia do Paraná (TECPAR), Curitiba, Paraná
  - Hospital Universitário Pedro Ernesto/ UERJ, Rio de Janeiro
  - Policlinica Lincoln de Freitas Filho, Rio de Janeiro
  - Unidade de Ensaios Clínicos em Imunobiológicos, Rio de Janeiro